CLINICAL TRIAL: NCT02423343
Title: A Phase 1b/2 Dose Escalation and Cohort Expansion Study of the Safety, Tolerability and Efficacy of a Novel Transforming Growth Factor-beta Receptor I Kinase Inhibitor (Galunisertib) Administered in Combination With Anti-PD-1 (Nivolumab) in Advanced Refractory Solid Tumors (Phase 1b) and in Recurrent or Refractory Non-small Cell Lung Cancer or Hepatocellular Carcinoma (Phase 2)
Brief Title: A Study of Galunisertib (LY2157299) in Combination With Nivolumab in Advanced Refractory Solid Tumors and in Recurrent or Refractory NSCLC, or Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15702; H9H-MC-JBEF (Other: Eli Lilly and Company); 2015-002093-20 (EudraCT Number)
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Solid Tumor; Non-Small Cell Lung Cancer Recurrent; Hepatocellular Carcinoma Recurrent
MeSH Terms: interventions — LY-2157299; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Galunisertib + Nivolumab (Cohort 1) Phase 1b (Experimental): 50 milligrams (mg) Galunisertib administered orally once daily (QD) on Day 1 through Day 14 of each 4-week cycle in combination with 3 milligrams per kilogram (3 mg/kg) nivolumab given intravenously (IV), every 2 weeks (Q2W), (Day 1 and Day 15). Participants may continue to receive study drug until discontinuation criteria are met.
  Interventions: Drug: Galunisertib; Drug: Nivolumab
- Galunisertib + Nivolumab (Cohort 2) Phase 1b (Experimental): 50 mg Galunisertib administered orally twice daily (BID) on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV, Q2W,(Day 1 and Day 15). Participants may continue to receive study drug until discontinuation criteria are met.
  Interventions: Drug: Galunisertib; Drug: Nivolumab
- Galunisertib + Nivolumab (Cohort 3) Phase 1b (Experimental): 80 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV, Q2W, (Day 1 and Day 15). Participants may continue to receive study drug until discontinuation criteria are met.
  Interventions: Drug: Galunisertib; Drug: Nivolumab
- Galunisertib + Nivolumab (Cohort 4) Phase 1b (Experimental): 150 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV, Q2W,(Day 1 and Day 15). Participants may continue to receive study drug until discontinuation criteria are met.
  Interventions: Drug: Galunisertib; Drug: Nivolumab
- Galunisertib + Nivolumab - Non-small Cell Lung Cancer (NSCLC) Phase 2 (Experimental): 150 mg Galunisertib administered orally BID for the first 14 days of each 4-week cycle in combination with 3 mg/kg nivolumab given IV, Q2W, (Day 1 and Day 15) of each 4-week cycle. Participants may continue to receive study drug until discontinuation criteria are met.
  Interventions: Drug: Galunisertib; Drug: Nivolumab
- Galunisertib + Nivolumab - Hepatocellular Carcinoma (HCC) Phase 2 (Experimental): 150 mg Galunisertib administered orally BID for the first 14 days of each 4-week cycle in combination with 3 mg/kg nivolumab given IV, Q2W, (Day 1 and Day 15) of each 4-week cycle. Participants may continue to receive study drug until discontinuation criteria are met.
  Interventions: Drug: Galunisertib; Drug: Nivolumab

INTERVENTIONS:
Drug: Galunisertib — Administered orally
  Other Names: LY2157299
Drug: Nivolumab — Administered IV
  Other Names: OPDIVO®

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, and efficacy of the study drug known as galunisertib in combination with nivolumab in participants with advanced refractory solid tumors and in recurrent or refractory non-small cell lung cancer (NSCLC) or hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* For Phase 1b, must have advanced refractory solid tumors in any line of therapy.
* For Phase 2, must have one of the following tumor types: recurrent or refractory NSCLC (any histology), or HCC with elevated alpha-fetoprotein (AFP) ≥200 nanogram/milliliter (ng/mL).
* For Phase 2 only, have had disease progression or be refractory or intolerant to 1 prior line of therapy (first line therapy) for recurrent or refractory for NSCLC or HCC and have refused currently approved second-line therapy. First line therapy is defined as therapy used to treat advanced disease. This may include multiple chemotherapeutic, targeted or immunotherapeutic agents with or without radiation therapy and/or surgery. Each subsequent line of therapy is preceded by disease progression. A switch of an agent within the same drug class (eg, cisplatinum to carboplatinum) within a regimen in order to manage toxicity does not define the start of a new line of therapy.
* For NSCLC:

  * Prior lines of therapy must include a platinum-based therapy. Investigational agents used in combination with standard therapies are allowed. Participants who received platinum-based neoadjuvant or adjuvant therapy and subsequently received platinum-based therapy as first-line therapy are eligible.
  * Participants who have completed neo-adjuvant or adjuvant therapy with a platinum doublet and have experienced disease recurrence within 6 months of completing the platinum doublet are eligible.
  * Tumors with driver mutations (epidermal growth factor receptor mutation positive or anaplastic lymphoma kinase fusion oncogene positive) treated with a tyrosine kinase inhibitor or crizotinib are eligible. For participants who have progressed on a tyrosine kinase inhibitor or crizotinib or are intolerant to this targeted therapy, that participant must receive platinum-based therapy prior to enrollment in this study. Documentation of such mutations must be available and entered into the electronic case report form (eCRF).
  * Maintenance or switch maintenance therapy after first-line chemotherapy will be considered part of the first-line regimen and is acceptable.

Participants who completed and progressed on a platinum-containing regimen as adjuvant, neoadjuvant, or part of a course of chemoradiation therapy given from locally advanced disease and developed recurrent (local or metastatic) disease within the 6 months before screening would be counted as having received 1 prior platinum-containing regimen and therefore would not require re-treatment with a platinum-containing regimen for Stage IIIB, IV, or recurrent disease and are eligible. However, participants must have received at least 2 cycles of a platinum doublet based chemotherapy before discontinuation for toxicity. If participants received only one cycle of a platinum doublet and discontinue due to clear progression, that regimen should be counted as a prior line of therapy.

* For HCC:

  * One prior line of therapy which must include sorafenib or participant must have progressed or been intolerant to sorafenib for participants not eligible for transarterial chemoembolization. Participants who had sorafenib for locally advanced disease or are intolerant to sorafenib are eligible. Participants may have had clinical progression only following sorafenib or local therapy.
  * Must have Child-Pugh A only. Participants may have any viral status (hepatitis B, hepatitis C, or none).
  * Have a viral load <100 international units/milliliter (IU/mL).
  * For hepatitis B participants, must be on a nucleoside analog reverse transcriptase inhibitor (lamivudine, telbivudine, adefovir, tenofovir, or entecavir).
* Have adequate organ function.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Use an approved contraceptive method.

Exclusion Criteria:

* For Phase 2 only, more than 1 prior line of therapy for their tumor type.
* Have moderate or severe cardiovascular disease:

  * Have the presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension.
  * Have documented major electrocardiogram (ECG) abnormalities which are clinically significant at the investigator's discretion (for example, symptomatic or sustained atrial or ventricular arrhythmias, second- or third-degree atrioventricular block, bundle-branch blocks, ventricular hypertrophy, or recent myocardial infarction).
  * Have major abnormalities documented by ECHO with Doppler:
  * Moderate or severe heart valve function defect including moderate or severe valve stenosis or regurgitation.
  * Left ventricular (LV) ejection fraction <50%, evaluation based on the institutional lower limit of normal.
  * Have septal aneurysm or other heart aneurysm.
  * Any aneurysm of the major vessels.
* Active infection with hepatitis B virus (HBV) (positive hepatitis B surface antigen); HCV is allowed only in HCC participants. HCC participants at risk for HBV reactivation (as defined by anti-hepatitis B core antibody positive) are only eligible in the HCC cohort.
* Have evidence of interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity or active, noninfectious pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (5):
  - University of Alabama at Birmingham Medical Center, Birmingham, Alabama
  - University of California - San Diego, La Jolla, California
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga, Málaga

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Nadal E, Saleh M, Aix SP, Ochoa-de-Olza M, Patel SP, Antonia S, Zhao Y, Gueorguieva I, Man M, Estrem ST, Liu J, Avsar E, Lin WH, Benhadji KA, Gandhi L, Guba SC, Diaz IA. A phase Ib/II study of galunisertib in combination with nivolumab in solid tumors and non-small cell lung cancer. BMC Cancer. 2023 Jul 28;23(1):708. doi: 10.1186/s12885-023-11153-1. PMID 37507657
- See also: Description: Click here for more information about this study: A Study of Galunisertib (LY2157299) in Combination With Nivolumab in Advanced Refractory Solid Tumors and in Recurrent or Refractory NSCLC, or Hepatocellular Carcinoma. — http://www.lillytrialguide.com/en-US/studies/solid-tumor/JBEF#?postal=jbef

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due low enrollment, the Hepatocellular Carcinoma (HCC) cohort was terminated early.
Pre-assignment Details: Participants who had at least one post baseline tumor assessment were considered to have completed the study.
Groups:
- Galunisertib + Nivolumab (Cohort 1) Phase 1b: 50 milligram (mg) Galunisertib administered orally daily (QD) on Day 1 through Day 14 of each 4-week cycle in combination with 3 milligrams per kilogram (3 mg/kg) nivolumab given intravenously (IV), every 2 weeks (Q2W), on Day 1 and Day 15 for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 2) Phase 1b: 50 mg Galunisertib administered orally twice daily (BID) on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV, Q2W, on Day 1 and Day 15 for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 3) Phase 1b: 80 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV, Q2W, on Day 1 and Day 15 for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 4) Phase 1b: 150 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV, Q2W, on Day 1 and Day 15 for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab - Non-Small Cell Lung Cancer (NSCLC) Phase 2; Galunisertib + Nivolumab - Hepatocellular Carcinoma (HCC) Phase 2: 150 mg Galunisertib administered orally BID for the first 14 days of each 4 week cycle in combination with 3 mg/kg nivolumab given IV, Q2W, (Day 1 and Day 15) of each 4-week cycle. Participants may continue to receive study drug until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Galunisertib + Nivolumab (Cohort 1) Phase 1b | Galunisertib + Nivolumab (Cohort 2) Phase 1b | Galunisertib + Nivolumab (Cohort 3) Phase 1b | Galunisertib + Nivolumab (Cohort 4) Phase 1b | Galunisertib + Nivolumab - Non-Small Cell Lung Cancer (NSCLC) Phase 2 | Galunisertib + Nivolumab - Hepatocellular Carcinoma (HCC) Phase 2
Started | 3 | 5 | 3 | 4 | 25 | 1
Received at Least One Dose of Study Drug | 3 | 5 | 3 | 4 | 25 | 1
Completed | 3 | 4 | 3 | 4 | 20 | 1
Not Completed | 0 | 1 | 0 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Galunisertib + Nivolumab (Cohort 1) Phase 1b: 50 mg Galunisertib administered orally daily on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given intravenously (IV) every 2 weeks (Day 1 and Day 15) for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 2) Phase 1b: 50 mg Galunisertib administered orally twice daily on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV every 2 weeks (Day 1 and Day 15) for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 3) Phase 1b: 80 mg Galunisertib administered orally twice daily on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV every 2 weeks(Day 1 and Day 15) for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 4) Phase 1b: 150 mg Galunisertib administered orally twice daily on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV every 2 weeks (Day 1 and Day 15) for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab - Non Small Cell Lung Cancer (NSCLC) Phase 2; Galunisertib + Nivolumab - Hepatocellular Carcinoma(HCC) Phase 2: 150 mg Galunisertib given orally twice daily for the first 14 days of each 4 week cycle in combination with 3 mg/kg nivolumab given IV every 2 weeks (Day 1 and Day 15) of each 4-week cycle. Participants may continue to receive study drug until discontinuation criteria are met.
- Total: Total of all reporting groups
Arm/Group | Galunisertib + Nivolumab (Cohort 1) Phase 1b | Galunisertib + Nivolumab (Cohort 2) Phase 1b | Galunisertib + Nivolumab (Cohort 3) Phase 1b | Galunisertib + Nivolumab (Cohort 4) Phase 1b | Galunisertib + Nivolumab - Non Small Cell Lung Cancer (NSCLC) Phase 2 | Galunisertib + Nivolumab - Hepatocellular Carcinoma(HCC) Phase 2 | Total
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 25 | 1 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (15.6) | 47.2 (15.8) | 36.0 (5.3) | 61.5 (9.0) | 61.0 (8.4) | 64.0 (NA) — N =1 mean (SD) not available, individual value reported. | 57.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3 | 9 | 1 | 16
  Male | 2 | 4 | 2 | 1 | 16 | 0 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 2
  White | 2 | 5 | 3 | 3 | 25 | 1 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 2 | 4 | 1 | 0 | 13
  Spain | 0 | 2 | 1 | 0 | 24 | 1 | 28

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Maximum Tolerated Dose (MTD) of Galunisertib in Combination With Nivolumab
Description: The MTD is defined as the highest tested dose that has less than 33% probability of causing a dose limiting toxicity (DLT).
Time Frame: Cycle 1 through Cycle 2 (Up to 2 Months)
Population: All participants who received at least one dose of study drug in Phase 1b per protocol.
Measure: Number; unit: milligrams (mg)
Groups:
- Phase 1b Participants: Cohort 1: 50 mg Galunisertib administered QD on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV, every Q2W, on Day 1 and Day 15 for 2 cycles.
  Cohort 2: 50 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W on Day 1 and Day 15 for 2 cycles.
  Cohort 3: 80 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W on Day 1 and Day 15 for 2 cycles.
  Cohort 4: 150 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W on Day 1 and Day 15 for 2 cycles.
Arm/Group | Phase 1b Participants
Number analyzed (Participants) | 15
milligrams (mg) | 300

2. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Nivolumab
Description: Minimum Concentration (Cmin) of Nivolumab
Time Frame: PK: Cycle 1 Day 15 Predose; Cycle 2: Day 1: Pre-dose; Day 15: Predose: Cycle 4: Day 1: Predose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Full Range); unit: micrograms per milliliter (µg/mL)
Groups:
- Galunisertib + Nivolumab (Cohort 1) Phase 1b: 50 mg Galunisertib administered orally QD on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV every Q2W on Day 1 and Day 15 for 2 cycles.
- Galunisertib + Nivolumab (Cohort 2) Phase 1b: 50 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W on Day 1 and Day 15 for 2 cycles.
- Galunisertib + Nivolumab (Cohort 3) Phase 1b: 80 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W on Day 1 and Day 15 for 2 cycles.
- Galunisertib + Nivolumab (Cohort 4) Phase 1b: 150 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W on Day 1 and Day 15 for 2 cycles.
- Galunisertib + Nivolumab (NSCLC) Phase 2; Galunisertib + Nivolumab ( HCC) Phase 2: 150 mg Galunisertib administered orally BID for the first 14 days of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W (Day 1 and Day 15) of each 4-week cycle. Participants may continue to receive study drug until discontinuation criteria are met.
Arm/Group | Galunisertib + Nivolumab (Cohort 1) Phase 1b | Galunisertib + Nivolumab (Cohort 2) Phase 1b | Galunisertib + Nivolumab (Cohort 3) Phase 1b | Galunisertib + Nivolumab (Cohort 4) Phase 1b | Galunisertib + Nivolumab (NSCLC) Phase 2 | Galunisertib + Nivolumab ( HCC) Phase 2
Number analyzed (Participants) | 2 | 5 | 3 | 4 | 11 | 0
micrograms per milliliter (µg/mL) | 33.5 [19.9 to 53.6] | 36.2 [11.8 to 58.1] | 43.2 [5.45 to 76] | 29.2 [9.39 to 63.7] | 37.6 [1.08 to 105] |

3. Secondary Outcome: PK: Area Under the Plasma Concentration -Time Curve of Galunisertib From Time Zero to 24 Hours (AUC [0-24h]) at Steady State
Description: Area under the plasma concentration curve from time zero to 24 hours of galunisertib for Cycle 1 and Cycle 2.
Time Frame: PK: Cycle 1 and Cycle 2 Day 1: Predose, 0.5 - 3 hours postdose, Cycle 1 and Cycle 2 Day 14: Predose, 0.5 - 2, 3.5 - 5, and 24 hours postdose through Cycle 4 Day 1 predose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per liter (μg*h/L)
Groups:
- Galunisertib + Nivolumab (Cohort 1) Phase 1b: 50 mg Galunisertib administered orally QD on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W (Day 1 and Day 15) for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 2) Phase 1b: 50 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W (Day 1 and Day 15) for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 3) Phase 1b: 80 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W (Day 1 and Day 15) for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 4) Phase 1b: 150 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W (Day 1 and Day 15) for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (NSCLC ) Phase 2; Galunisertib + Nivolumab ( HCC) Phase 2: 150 mg Galunisertib administered orally BID for the first 14 days of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W (Day 1 and Day 15) of each 4-week cycle. Participants may continue to receive study drug until discontinuation criteria are met.
Arm/Group | Galunisertib + Nivolumab (Cohort 1) Phase 1b | Galunisertib + Nivolumab (Cohort 2) Phase 1b | Galunisertib + Nivolumab (Cohort 3) Phase 1b | Galunisertib + Nivolumab (Cohort 4) Phase 1b | Galunisertib + Nivolumab (NSCLC ) Phase 2 | Galunisertib + Nivolumab ( HCC) Phase 2
Number analyzed (Participants) | 3 | 4 | 3 | 4 | 12 | 1
micrograms*hour per liter (μg*h/L) | 3060 (41) | 2350 (46) | 2220 (164) | 5580 (61) | 7322 (67) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there was only one participant. Individual value reported: 6005 μg*h/L

4. Secondary Outcome: Number of Participants With Anti-Nivolumab Antibodies When Administered in Combination With Galunisertib
Description: Participants with treatment-emergent anti-nivolumab antibodies when administered with galunisertib were participants with a 4-fold or greater increase in titer from baseline measurement (treatment-boosted). If baseline result is ADA not present, then the subject is TE ADA+, if there is at least 1 postbaseline result of ADA present with titer ≥ 40 (treatment-induced).
Time Frame: Cycle 1: Days 1, 14, 15 Predose and Day 100 Follow-up; Cycles 2 and 4: Day 1 Predose and Day 100 Follow-up
Population: All participants who received at least one dose of study drug and were evaluable for TE ADA.
Measure: Count of Participants; unit: Participants
Groups:
- Galunisertib + Nivolumab (Cohort 1) Phase 1b: 50 mg Galunisertib administered orally QD on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV every Q2W on Day 1 and Day 15 for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 2) Phase 1b: 50 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W on Day 1 and Day 15 for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 3) Phase 1b: 80 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W on Day 1 and Day 15 for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (Cohort 4) Phase 1b: 150 mg Galunisertib administered orally BID on Day 1 through Day 14 of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W on Day 1 and Day 15 for 2 cycles. Participants may continue to receive study drug until discontinuation criteria are met.
- Galunisertib + Nivolumab (HCC) Phase 2: 150 mg Galunisertib administered orally BID for the first 14 days of each 4-week cycle in combination with 3 mg/kg nivolumab given IV Q2W (Day 1 and Day 15) of each 4-week cycle. Participants may continue to receive study drug until discontinuation criteria are met.
Arm/Group | Galunisertib + Nivolumab (Cohort 1) Phase 1b | Galunisertib + Nivolumab (Cohort 2) Phase 1b | Galunisertib + Nivolumab (Cohort 3) Phase 1b | Galunisertib + Nivolumab (Cohort 4) Phase 1b | Galunisertib + Nivolumab (NSCLC) Phase 2 | Galunisertib + Nivolumab (HCC) Phase 2
Number analyzed (Participants) | 3 | 5 | 2 | 3 | 13 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of first study treatment to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: Date of First Study Treatment to Measured Progressive Disease or Death (Up to 35 Months)
Population: All participants who received at least one dose of study drug in the Phase 2 cohorts. Censored participants Galunisertib + Nivolumab (NSCLC) Phase 2 = 6.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Galunisertib + Nivolumab (NSCLC) Phase 2 | Galunisertib + Nivolumab (HCC) Phase 2
Number analyzed (Participants) | 25 | 1
months | 5.26 [1.77 to 9.20] | 5.39

6. Secondary Outcome: Phase 2: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response or Partial Response: Objective Response Rate (ORR)
Description: Objective Response Rate was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Baseline to Measured Progressive Disease (Up to 35 Months)
Population: All participants who received at least one dose of study drug in Phase 2 cohorts.
Measure: Number; unit: Percentage of Participants
Arm/Group | Galunisertib + Nivolumab (NSCLC) Phase 2 | Galunisertib + Nivolumab (HCC) Phase 2
Number analyzed (Participants) | 25 | 1
Percentage of Participants | 24.0 | 0

7. Secondary Outcome: Phase 2: Duration of Response (DoR)
Description: Duration of response was measured from the date of documented response to the date of first progression of disease or the date of death due to any cause, whichever is earlier.
Time Frame: Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression or Death Due to Any Cause (Up to 35 Months)
Population: All participants who received at least one dose of study drug in Phase 2 cohorts and had a response of complete response or partial response. Censored participants Galunisertib + Nivolumab (NSCLC) Phase 2 = 1.
Measure: Median (Full Range); unit: months
Groups:
- Galunisertib + Nivolumab (HCC) Phase 2: 150 mg Galunisertib administered orally BID for the first 14 days of each 4-week cycle in combination with 3 mg/kg nivolumab given IV every 2 weeks (Day 1 and Day 15) of each 4-week cycle. Participants may continue to receive study drug until discontinuation criteria are met.
Arm/Group | Galunisertib + Nivolumab (NSCLC) Phase 2 | Galunisertib + Nivolumab (HCC) Phase 2
Number analyzed (Participants) | 6 | 0
months | 9.03 [1.97 to 35] |

8. Secondary Outcome: Phase 2: Time to Response
Description: Time to response was measured from the date of first study treatment to the first documented response of Complete Response (CR) or Partial Response (PR).
Time Frame: Date of First Study Treatment to Date of Complete Response or Partial Response (Up to 35 Months)
Population: All participants who received at least one dose of study drug in Phase 2 cohorts and had a documented response of CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | Galunisertib + Nivolumab (NSCLC) Phase 2 | Galunisertib + Nivolumab (HCC) Phase 2
Number analyzed (Participants) | 6 | 0
months | 4.2 [0.5 to 35] |

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: Overall Survival was determined from the date of first study treatment until death due to any cause.
Time Frame: Date of First Study Treatment to Death from Any Cause (Up to 35 Months)
Population: All participants who received at least one dose of study drug in Phase 2 cohorts. Censored participants Galunisertib + Nivolumab (NSCLC) Phase 2 = 8.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Galunisertib + Nivolumab (NSCLC) Phase 2 | Galunisertib + Nivolumab (HCC) Phase 2
Number analyzed (Participants) | 25 | 1
months | 11.99 [8.15 to 16.23] | 14.52

ADVERSE EVENTS:
Time Frame: Up to 35 months
Description: All participants who received at least one dose of study drug.
Arm/Group | Galunisertib + Nivolumab (Cohort 1) Phase 1b | Galunisertib + Nivolumab (Cohort 2) Phase 1b | Galunisertib + Nivolumab (Cohort 3) Phase 1b | Galunisertib + Nivolumab (Cohort 4) Phase 1b | Galunisertib + Nivolumab (NSCLC) Phase 2 | Galunisertib + Nivolumab (HCC) Phase 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/5 | 1/3 | 3/4 | 17/25 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/5 | 1/3 | 2/4 | 13/25 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 4/5 | 3/3 | 4/4 | 23/25 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galunisertib + Nivolumab (Cohort 1) Phase 1b (N=3) | Galunisertib + Nivolumab (Cohort 2) Phase 1b (N=5) | Galunisertib + Nivolumab (Cohort 3) Phase 1b (N=3) | Galunisertib + Nivolumab (Cohort 4) Phase 1b (N=4) | Galunisertib + Nivolumab (NSCLC) Phase 2 (N=25) | Galunisertib + Nivolumab (HCC) Phase 2 (N=1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Noninfective encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galunisertib + Nivolumab (Cohort 1) Phase 1b (N=3) | Galunisertib + Nivolumab (Cohort 2) Phase 1b (N=5) | Galunisertib + Nivolumab (Cohort 3) Phase 1b (N=3) | Galunisertib + Nivolumab (Cohort 4) Phase 1b (N=4) | Galunisertib + Nivolumab (NSCLC) Phase 2 (N=25) | Galunisertib + Nivolumab (HCC) Phase 2 (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (3) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (5) | 0 (0) | 1 (1) | 7 (10) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 6 (6) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 6 (10) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (4) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (4) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cd4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystatin c increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Troponin t increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (11) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (6) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neurological symptom (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 9 (14) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (10) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due low enrollment, the HCC cohort was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/43/NCT02423343/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT02423343/SAP_001.pdf